CLINICAL TRIAL: NCT00874770
Title: A Phase 2a Study of BMS-790052 in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Treatment Naive Subjects With Chronic Hepatitis C Virus Genotype 1
Brief Title: Safety and Efficacy of Daclatasvir (BMS-790052) Plus Standard of Care (Pegylated-interferon Alpha and Ribavirin)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI444-014; EUDRACT# 2009-010149-29
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Infection
Keywords: Antivirals
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Daclatasvir, plus Peginterferon alpha-2a, ribavirin (A) (Experimental): Active Comparator
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alpha-2a; Drug: ribavirin
- Daclatasvir, Peginterferon alpha-2a, ribavirin (B) (Experimental): Active Comparator
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alpha-2a; Drug: ribavirin
- Daclatasvir, Peginterferon alpha-2a, ribavirin (C) (Experimental): Active Comparator
  Interventions: Drug: Daclatasvir; Drug: Peginterferon alpha-2a; Drug: ribavirin
- Placebo, Peginterferon alpha-2a, ribavirin (D) (Active Comparator)
  Interventions: Drug: Placebo; Drug: Peginterferon alpha-2a; Drug: ribavirin

INTERVENTIONS:
Drug: Daclatasvir — Tablets, oral, 3 mg, Daily, 48 weeks
  Arms: Daclatasvir, plus Peginterferon alpha-2a, ribavirin (A)
Drug: Daclatasvir — Tablets, oral, 10 mg, Daily, 48 weeks
  Arms: Daclatasvir, Peginterferon alpha-2a, ribavirin (B)
Drug: Daclatasvir — Tablets, oral, 60 mg, Daily, 48 weeks
  Arms: Daclatasvir, Peginterferon alpha-2a, ribavirin (C)
Drug: Placebo — Tablet, oral, 0 mg, Daily 48 weeks
  Arms: Placebo, Peginterferon alpha-2a, ribavirin (D)
Drug: Peginterferon alpha-2a — Syringe, subcutaneous, 180 µg, Weekly, 48 weeks
  Other Names: Pegasys
Drug: ribavirin — Tablet, oral, 1000 or 1200 mg, based on weight, Daily, 48 weeks
  Other Names: Copegus

SUMMARY:
The purpose of this study is to identify 1 or more doses of daclatasvir, which when used in combination with pegylated interferon alpha and ribavirin, are safe and demonstrate sufficient anti-hepatitis C virus activity.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients chronically infected with hepatitis C virus (HCV) genotype 1
* HCV RNA viral load of ≥10*5* IU/mL (100,000 IU/mL) at screening
* Treatment naive

Key Exclusion Criteria:

* Women of child-bearing potential
* Cirrhosis
* Coinfection with HIV or hepatitis B virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (11):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Mercy Medical Center, Baltimore, Maryland
  - Llc Dba The Research Institute, Springfield, Massachusetts
  - Veterans Affairs Medical Center, The Bronx, New York
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - North Texas Research Institute, Arlington, Texas
  - Metropolitan Research, Fairfax, Virginia
- France (3):
  - Local Institution, Créteil
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Pol S, Ghalib RH, Rustgi VK, Martorell C, Everson GT, Tatum HA, Hezode C, Lim JK, Bronowicki JP, Abrams GA, Brau N, Morris DW, Thuluvath PJ, Reindollar RW, Yin PD, Diva U, Hindes R, McPhee F, Hernandez D, Wind-Rotolo M, Hughes EA, Schnittman S. Daclatasvir for previously untreated chronic hepatitis C genotype-1 infection: a randomised, parallel-group, double-blind, placebo-controlled, dose-finding, phase 2a trial. Lancet Infect Dis. 2012 Sep;12(9):671-7. doi: 10.1016/S1473-3099(12)70138-X. Epub 2012 Jun 18. PMID 22714001
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in France and USA.
Pre-assignment Details: A total of 74 participants were enrolled, of which 48 were randomized to receive treatment and 26 were not randomized: 22 no longer met study criteria, 2 withdrew consent, 1 was lost to follow-up, and 1 due to other reasons.
Groups:
- Daclatasvir 3 mg + pegIFNα-2a + Ribavirin: Participants received 3 mg of daclatasvir once daily (OD) in coadministration with peginterferon alpha-2a (pegIFNα-2a)180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10 mg of daclatasvir OD coadministered with pegIFNα-2a 180 µg given subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 60 mg + pegIFNα-2a + Ribavirin: Participants received 60 mg of daclatasvir OD in coadministration with pegIFNα-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Placebo+pegIFNα-2a+Ribavirin: Participants received a matching placebo of daclatasvir tablets administered orally once daily for 48 weeks in coadministration with pegIFNα-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Period: Overall Study
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo+pegIFNα-2a+Ribavirin
Started | 12 | 12 | 12 | 12
Completed | 7 | 11 | 8 | 7
Not Completed | 5 | 1 | 4 | 5
Not completed — Lack of Efficacy | 2 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Subject no Longer Meets Study Criteria | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed in the treated population defined as all participants who received at least 1 dose of study therapy.
Groups:
- Daclatasvir 3-mg+pegIFNα-2a-2a+Ribavirin: Participants received 3 mg of daclatasvir once daily (OD) in coadministration with peginterferon alpha-2a (pegIFNα-2a)180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 10-mg+pegIFNα-2a+Ribavirin: Participants received 10-mg of daclatasvir OD in coadministration with pegIFNα-2a-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 60-mg+pegIFNα-2a+Ribavirin: Participants received 60-mg of daclatasvir OD in coadministration with pegIFNα-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Total: Total of all reporting groups
Arm/Group | Daclatasvir 3-mg+pegIFNα-2a-2a+Ribavirin | Daclatasvir 10-mg+pegIFNα-2a+Ribavirin | Daclatasvir 60-mg+pegIFNα-2a+Ribavirin | Placebo+pegIFNα-2a+Ribavirin | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8.56) | 53.2 (9.11) | 52 (7.34) | 48 (10.20) | 51.3 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 4 | 16
  Male | 9 | 8 | 7 | 8 | 32

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), and Treatment-related AEs and Who Died in Treatment Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a patient or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Treatment-related AE was defined as an AE that had certain, probable, possible, or unknown relationship to study drug.
Time Frame: SAE: From Day 1 up to 30 days after last dose of study drug, AE: From Day 1 to 7 days after last dose of study drug
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Daclatasvir 3 mg + pegIFNα-2a + Ribavirin: Participants received 3 mg of daclatasvir once daily (OD) coadministered orally with peginterferon alpha-2a (pegIFNα-2a)180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10 mg of daclatasvir OD coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 60 mg + pegIFNα-2a + Ribavirin: Participants received 60 mg of daclatasvir OD coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Placebo + pegIFNα-2a + Ribavirin: Participants received a matching placebo of daclatasvir tablets coadministered orally once daily for 48 weeks with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
participants
  SAEs | 1 | 1 | 1 | 0
  Discontinuation due to AEs | 1 | 1 | 4 | 2
  Grade 2 to 4 Related AEs | 6 | 6 | 9 | 7
  Deaths | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), and Treatment-related AEs and Who Died in Follow-up Period
Description: as for outcome 1
Time Frame: From Day 31 up to Week 24 of post treatment follow-up
Population: All participants who received at least 1 dose of study drug. n=evaluable patients
Measure: Number; unit: participants
Groups:
- Daclatasvir 3 mg + pegIFNα-2a + Rribavirin: Participants received 3 mg of daclatasvir once daily (OD) coadministered orally with peginterferon alpha-2a (pegIFNα-2a)180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Rribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
participants
  SAEs (n=10,12,12,10) | 0 | 0 | 3 | 0
  Discontinuation due to AEs | 0 | 0 | 0 | 0
  Grade 2 to 4 Related AEs | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR) at Weeks 4 and 12
Description: eRVR was defined as undetectable hepatitis C virus RNA less than the lower limit of detection (10 IU/mL) at Weeks 4 and 12.
Time Frame: A Weeks 4 and 12
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Daclatasvir 60 mg + pegIFNα-2a + Ribavirin: Participants received 60 mg of daclatasvir OD in coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants | 41.7 | 83.3 | 75 | 8.3

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR) at Week 4
Description: RVR was defined as undetectable hepatitis C virus (HCV) RNA ie, HCV RNA less than the lower limit of detection (10 IU/mL) at Week 4.
Time Frame: At Week 4
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10-mg of daclatasvir OD coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Placebo + pegIFNα-2a + Ribavirin: Participants received a matching placebo of daclatasvir tablets coadministered orally once daily for 48 weekswith pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants | 41.7 | 91.7 | 83.3 | 8.3

5. Secondary Outcome: Percentage of Participants With Early Virologic Response (EVR) at Week 12
Description: EVR was defined as a ≥2 log10 decrease in hepatitis C virus (HCV) RNA from baseline at Week 12 , or HCV RNA <10 IU/mL for participants with baseline HCV RNA <1000 IU/mL.
Time Frame: At Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10 mg of daclatasvir OD in coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants | 75 | 100 | 83.3 | 66.7

6. Secondary Outcome: Percentage of Participants With a Complete Early Virologic Response (cEVR) at Week 12
Description: cEVR was defined as hepatitis C virus RNA <10 IU/mL at Week 12
Time Frame: At Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Daclatasvir 3 mg + pegIFNα-2a + Riibavirin: Participants received 3 mg of daclatasvir once daily (OD) coadministered orally with peginterferon alpha-2a (pegIFNα-2a)180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10 mg of daclatasvir OD coadministered orally with pegIFNα-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 60 mg + pegIFNα-2a + Ribavirin: Participants received 60 mg of daclatasvir OD coadministered orally with pegIFNα-2a 180 µg administered subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Placebo + pegIFNα-2a + Ribavirin: Participants received a matching placebo of daclatasvir tablets coadministered orally once daily for 48 weeks with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).48 weeks.
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Riibavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants | 58.3 | 83.3 | 83.3 | 41.7

7. Other Pre Specified Outcome: Number of Participants With Grade 3 to 4 Abnormalities on Laboratory Test Results
Description: Clinically significant change in marked laboratory abnormalities (Grade 3 to 4 ) included: Alanine aminotransferase (ALT)- Grade 3 as >5.0 to 10.0* Upper Limit of Normal (ULN), Grade 4 as >10.0*ULN; Aspartate aminotransferase (AST)- Grade 3 as >5.0 to 10.0*ULN, Grade 4 as >10.0*ULN; Hemoglobin- Grade 3 as 7.0 to 8.9 g/dL, Grade 4 as <7.0 g/dL; Neutrophils- Grade 3 as 0.5 to 0.749*10^9/L, Grade 4 as <0.5*10^9/L; Lymphocytes- Grade 3 as 0.35 to 0.499*10^9/L, Grade 4 as <0.35*10^9/L; Total Bilirubin- Grade 3 as 2.6-5.0*ULN, Grade 4 as >5.0*ULN; Platelets- Grade 3 as 25000 to 49999*10^9/L, Grade 4 as <25000 10^9/L and white blood cells (WBC) - Grade 3 as 1000 to 1499*10^9/L, Grade 4 as <1000*10^9/L.
Time Frame: From screening up to Week 12 (treatment period)
Population: All participants who received at least 1 dose of study drug. n=evaluable patients at the specified time point
Measure: Number; unit: participants
Groups:
- Placebo + pegIFNα-2a + Ribavirin: Participants received a matching placebo of daclatasvir tablets once daily for 48 weeks coadministered orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Number analyzed (Participants) | 12 | 12 | 12 | 12
participants
  Hemoglobin (n= 11,12,12,11) | 1 | 0 | 1 | 0
  Lymphocytes (n= 11,12,12,12) | 1 | 3 | 3 | 3
  Neutrophils (n= 11,12,12,12) | 2 | 4 | 3 | 4
  Platelets (n= 11,12,12,12) | 0 | 0 | 0 | 1
  ALT (n= 11,12,12,12) | 0 | 1 | 0 | 3
  AST (n= 11,12,12,12) | 0 | 0 | 0 | 3
  Total bilirubin (n= 11,12,12,12) | 0 | 0 | 1 | 0
  WBC (n= 11, 12, 12, 12) | 0 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after last dose of drug
Groups:
- Daclatasvir 3 mg + pegIFNα-2a + Ribavirin: Participants received 3 mg of daclatasvir once daily (OD) in coadministration orally with peginterferon alpha-2a (pegIFNα-2a)180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 10 mg + pegIFNα-2a + Ribavirin: Participants received 10 mg of daclatasvir OD in coadministration orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Daclatasvir 60 mg + pegIFNα-2a + Ribavirin: Participants received 60 mg of daclatasvir OD in coadministration orally with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
- Placebo + pegIFNα-2a + Ribavirin: Participants received a matching placebo of daclatasvir tablets coadministered orally once daily for 48 weeks in with pegIFNα-2a 180 µg subcutaneously once weekly and ribavirin twice daily (400 mg tablets for participants <75 kg or 600 mg tablets for participants >75 kg in the morning with food and 600 mg tablets in the evening with food up to 48 weeks).
Arm/Group | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin | Placebo + pegIFNα-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin (N=12) | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin (N=12) | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin (N=12) | Placebo + pegIFNα-2a + Ribavirin (N=12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclatasvir 3 mg + pegIFNα-2a + Ribavirin (N=12) | Daclatasvir 10 mg + pegIFNα-2a + Ribavirin (N=12) | Daclatasvir 60 mg + pegIFNα-2a + Ribavirin (N=12) | Placebo + pegIFNα-2a + Ribavirin (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Blood pressure fluctuation (Vascular disorders) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 3 | 1 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0
Food aversion (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 1 | 0
Irritability (General disorders) | 3 | 6 | 3 | 2
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 4 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 3 | 1 | 5 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Fatigue (General disorders) | 6 | 7 | 6 | 9
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 3 | 6 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 4 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 3 | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 9 | 7 | 3 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Injection site irritation (General disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 4 | 5 | 6
Malaise (General disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 2 | 2
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 2 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2 | 3
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 3 | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 6 | 5
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 3
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 4 | 6
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Pain (General disorders) | 3 | 0 | 2 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single center publications until after disclosure of the clinical trial's primary publication.